CLINICAL TRIAL: NCT05424861
Title: Acupressure Application for Relief of Postpartum Uterine Pain During Breastfeeding: A Randomized Controlled Study
Brief Title: Nonpharmacological Method for Relief of Uterine Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Medipol University (Other)
Responsible Party: Principal Investigator, sena dilek, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek1
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Pain
Keywords: Pain; involution; breast-feeding
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Active Comparator): Postpartum 6-24 days in the acupressure group. Acupressure will be applied 1 time just before breastfeeding between hours. The visual analog scale, in which the introductory information form is filled by the researcher and the pain score is evaluated, will be marked by the participant once before breastfeeding, once at the 10th minute of breastfeeding, and once at the 20th minute, in total 3 times.
  Interventions: Behavioral: Acupressure group
- Control group (Active Comparator): Postpartum 6-24 days in the control group. Introductory information form will be filled by the researcher between hours. The visual analog scale, in which the pain score is evaluated, will be marked by the participant for a total of 3 times, once just before breastfeeding, once at the 10th minute of breastfeeding, and once at the 20th minute.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Acupressure group — A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position of the mother, leaving the application points open. The most preferred points LI4 and SP6 were selected among the points that were reported to be effective in relieving luterus pain by scanning the literature on the points to be compressed. Acupressure will be applied to the points (bidirectional, right and left) for 2 minutes, for a total of 8 minutes. Light pressure will be applied with the thumb of the practitioner's hand. Immediately after applying pressure for 2 minutes for each point, it is passed to the other point in the symmetrical region and the application is made without interruption. While practicing, the researcher will check the time using a digital wristwatch with a stopwatch.
  Arms: Acupressure group
Other: Control group — No application will be made. The mothers in this group will fill in the visual analog scale, which evaluates postpartum uterine pain 3 times between 6-24 hours after birth.
  Arms: Control group

SUMMARY:
Postpartum uterine pain is an important part of the postpartum period and is a concern for women, which can negatively affect maternal-neonatal attachment and breastfeeding. Acupressure allows midwives to make evidence-based independent practice in controlling postpartum uterine pain. The aim of this study is to determine the effectiveness of acupressure, which is a non-pharmacological intervention, for postpartum uterine pain after vaginal delivery. The research will be carried out between February 2022 and December 2022 with mothers who gave vaginal birth at Health Sciences University Kocaeli Derince Training and Research Hospital. The research will be carried out with two groups as acupressure and control groups. The sample number was calculated using the G*Power 3.1.9.2 program and the acupressure group: 61 and the control group: 61. It was planned to collect the research data with the Introductory Information Form and Visual Analog Scale in which Postpartum Uterine Pain was evaluated. Postpartum 6-24 days in the acupressure group. Acupressure will be applied once between hours, just before breastfeeding. The visual analog scale, in which the introductory information form is filled by the researcher and the pain score is evaluated, will be marked by the participant once before breastfeeding, once at the 10th minute of breastfeeding, and once at the 20th minute, in total 3 times. No application will be made to the control group. The data of the research will be evaluated using the Statistical Package 22.0 program for Social Sciences. In the evaluation of the data; descriptive statistics will be given as percentage, arithmetic mean±standard deviation, median and minimum-maximum values. Independent two-sample t-test will be used for normally distributed variables and Mann-Whitney U test will be used for non-normally distributed variables. Pearson Correlation test will be applied to determine the relationship between the pain intensity of the acupressure group and the tests and to determine the relationship between the tests. Statistical significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
Aim: The aim of our study is to determine the effectiveness of acupressure, which is a non-pharmacological intervention, for postpartum uterine pain after vaginal delivery.

Hypothesis(s):

H0: Acupressure application during breastfeeding after vaginal delivery has no effect on reducing uterine pain.

H1: Acupressure application during breastfeeding after vaginal delivery has an effect on reducing uterine pain.

Type of Research: This study was designed as a randomized controlled experimental study.

Research Universe: The universe of the research will be multiparous mothers who have given vaginal birth in the Alikahya Campus of Health Sciences University Kocaeli Derince Training and Research Hospital. In order to determine the sample size in the study, De Sousa et al. was calculated based on the study conducted by T.R. to examine the effect of transcutaneous electrical nerve stimulation on postpartum uterine contraction pain during breastfeeding. The sample size of the study was calculated using the G*Power 3.1.9.2 program and the mean and standard deviation values of the uterine contraction pain variable in the related article (De Sousa et al., 2014) were taken into account in calculating the effect size. The mean and standard deviation values of the uterine contraction pain variable in the experimental group were 3.56±1.78. In the control group, the mean and standard deviation values of the uterine contraction pain variable were 4.81±2.37. Using the mean and standard deviation values of the related article, the effect size was calculated as 0.5964125. The minimum number of individuals to be included in the sample of this study was calculated by taking G*Power 3.1.9.2 and effect size: 0.5964125, α= 0.05, power: 0.90, and the sample size was determined as at least 61 mothers in each group. (acupressure group: 61 and control group: 61). A total of 122 women were planned to be included in the study (Acupressure group: 61 women, control group: 61 women).

In which group the mothers included in the study will be, will be determined from the website of the random number generation program "Research Randomizer", and they will be divided into two groups. Thus, each mother's number and group number will be determined and recorded.

Data Collection Tools It is planned to collect the research data with the Introductory Information Form and the VAS, in which Postpartum Uterine Pain is evaluated.

Introductory Information Form: This form was created by researchers based on the literature. The form consists of a total of 24 questions questioning women's knowledge about socio-domographic, obstetric and breastfeeding-related variables.

VAS for Evaluation of Postpartum Uterine Pain: The patient marks his or her own pain on a 10 cm ruler, which is marked as "no pain" at one end and the most severe pain at the other end. The patient is told that there are two endpoints and to mark any place between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.

Application Procedure of the Research After obtaining the approval of the ethics committee and the permission of the institution, the mothers who had a vaginal birth in the last 24 hours and met the inclusion criteria of the study will be selected from the study, and those who do not comply will be excluded from the study. In the literature, uterine pain associated with breastfeeding is felt more intensely, especially after the first 6 hours after delivery, until the 48th hour. In addition, multiparas experience more pain than primiparas. In the hospital where we will study, women who have given birth normally stay for 24 hours and are discharged afterwards. Therefore, multiparous women between 6-24 hours after their vaginal delivery will be included in the study. Mothers who have given vaginal birth will be met between the first 6-24 hours after the birth. Participants will be informed that they can participate in the study without affecting the care received at the hospital and they can leave the study at any time, and their consent will be obtained. After participants are included in the study, they will be assigned to one of the study groups according to the electronic randomization table. The data will be filled in by the researcher in the Gynecology-3 service of the hospital by face-to-face interview, and the VAS for Evaluation of Postpartum Uterine Pain will be filled in by the women themselves.

VAS Evaluation of Postpartum Uterine Pain by mothers;

* Postpartum 6-24. 1 time just before breastfeeding between hours,
* 1 time in the 10th minute of breastfeeding,
* It will be filled 3 times in total, once at the 20th minute of breastfeeding. To mothers;
* Postpartum 6-24. Acupressure will not be applied to the acupressure group once between hours, and no application will be made to the control group.

Location: It is the point where the cambered muscle group is when the thumb and forefinger are brought closer together. In other words, it corresponds to the midpoint of the metacarpal bone of the index finger.

Application Technique: Press the point with the thumb/middle finger for 2 minutes in a circular or up and down direction along the meridian line. Work on 2 points on both legs separately or simultaneously.

Indications of the Point: Although this area is generally used for face, head and toothache, it is also a frequently preferred area to increase alertness and reduce fatigue.

Spleen Meridian 6th Point (Sanyinjiao/SP6):

Location: It is located on the inner side of the tibia, four fingers above the ankle.

Application Technique: Press the point with the thumb/middle finger for 2 minutes in a circular or up and down direction along the meridian line. Work on 2 points on both legs separately or simultaneously.

Indications of the Point: This point, which is generally used for urological and pelvic problems, menstrual pain and insomnia, is also preferred to reduce fatigue in various studies.

Acupressure Application Technique A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position for the mother, leaving the application points exposed. Among the points reported to have an effect on uterine pain for this study, acupressure application points are among the most preferred points in the literature, spleen meridian point 6 (SP6) and large intestine meridian 4 point (LI4), a total of 2 (from each point on both sides). : 4 points) detailed information about the point is given below. In addition, expert opinion was taken to determine the points.

Light pressure will be applied with the thumb of the practitioner's hand. Immediately after applying pressure for 2 minutes for each point, it will be moved to the other point in the symmetrical region and the application will be made without interruption. Although there is a difference in the order of use of the determined acupressure points, this study will be carried out symmetrically to the LI4 and SP6 points, respectively. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch.

Large Intestine Meridian 4th Point (He Gu/LI4):

Location: It is the point where the cambered muscle group is when the thumb and forefinger are brought closer together. In other words, it corresponds to the midpoint of the metacarpal bone of the index finger.

Application Technique: Press the point with the thumb/middle finger for 2 minutes in a circular or up and down direction along the meridian line. Work on 2 points on both legs separately or simultaneously.

Indications of the Point: Although this area is generally used for face, head and toothache, it is also a frequently preferred area to increase alertness and reduce fatigue.

Spleen Meridian 6th Point (Sanyinjiao/SP6):

Location: It is located on the inner side of the tibia, four fingers above the ankle.

Application Technique: Press the point with the thumb/middle finger for 2 minutes in a circular or up and down direction along the meridian line. Work on 2 points on both legs separately or simultaneously.

Indications of the Point: This point, which is generally used for urological and pelvic problems, menstrual pain and insomnia, is also preferred to reduce fatigue in various studies.

The data of the study will be evaluated using the Statistical Package for the Social Sciences (SPSS) 22.0 program. All data will first be evaluated with the Kolmogorov-Smirnov test for conformity to normal distribution, and then analyzed according to conformity to normal distribution. For descriptive statistics, percentages will be used in general, arithmetic mean±standard deviation for those suitable for normal distribution, median and minimum-maximum values for those that do not fit. Comparisons between groups for numerical variables of socio-demographic and clinical characteristics will be made with an independent two-sample t-test for normally distributed variables, and Mann-Whitney U test for non-normally distributed variables. Pearson Correlation test will be applied to determine the relationship between the fatigue severity of the experimental group and the tests and to determine the relationship between the tests. Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Having a single and live baby between 37-42 weeks of gestation,
* Normal spontaneous vaginal delivery,
* Multiparous,
* Having a baby weighing 2-4 kilograms,
* No general anesthetic agent was used at birth,
* Have not used a non-pharmacological method for pain before,
* Having a Visual Analogue Scale (VAS) score of 4 and above for uterine pain before breastfeeding,
* Not having breastfeeding problems,
* Not having any health problems (Tuberculosis, HIV, cancer, etc.),
* Having given birth at least 6 hours ago,
* Does not have any problems preventing communication,
* Able to read and write,
* Able to speak and understand Turkish,
* Volunteer mothers who agreed to participate in the study will be included.

Exclusion Criteria:

* Having a situation that prevents breastfeeding (galactosemia, congenital anomalies, etc.),
* Having postpartum complications (bleeding, infection, etc.),
* Separated from her baby for any reason after birth (in cases where the mother or baby is referred, hospitalized in intensive care or isolated),
* Having lost her baby,
* Having any complications during pregnancy (gestational diabetes, preeclampsia, Rh incompatibility, heart disease, etc.),
* With uterine anomaly,
* Tissue integrity deteriorated in the area to be treated,
* Taking painkillers in the last 6 hours,
* Smoking or using alcohol,
* Those with positive Covid-19 test will be excluded from the study. In addition, those who want to leave the research at any stage of the research will be excluded from the research.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 122 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for assessing postpartum uterine pain | This scale will be completed by the participants just before breastfeeding.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The patient is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.
Visual analog scale for assessing postpartum uterine pain | This scale will be completed by the participants at the 10th minute of breastfeeding.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The patient is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.
Visual analog scale for assessing postpartum uterine pain | This scale will be completed by the participants at the 20th minute of breastfeeding.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The patient is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D, Principal Investigator — Kocaeli University; Resmiye Kaya Odabas, MSc, Study Chair — Kocaeli University; Derya Kanza Gul, MD, Study Chair — Medipol University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No